CLINICAL TRIAL: NCT04552028
Title: Correlation of Non-invasive and Invasive Oxygenation for the Diagnosis of Respiratory Dysfunction in Acute Pancreatitis
Brief Title: Respiratory Dysfunction in Acute Pancreatitis (SAFI)
Acronym: SAFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. med. Hector Eloy Tamez Perez (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Hector Eloy Tamez Perez, Clinical Professor, Hospital Universitario Dr. Jose E. Gonzalez
Organization: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Other Study IDs: GA19-00011
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Acute Pancreatitis; Complication
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non invasive oxygenation — To determine if the SpO2 / FIO2 ratio has a correlation with PaO2 / FIO2 ratio to identify respiratory compromise in acute pancreatitis.

SUMMARY:
Acute pancreatitis (AP) is an inflammatory process of the pancreas and is one of the main causes of hospital admission of gastrointestinal origin. The annual incidence is between 13 to 45 per 100,000 habitants. The etiology may correspond to vesicular gallstones, excessive alcohol consumption, drugs, among others. Risk factors such as smoking and type 2 diabetes mellitus have been found to increase the risk of pancreatitis by 1.86 to 2.89 times.

Pulmonary complications are the most frequent in this group of patients, approximately in 75% of cases, they vary from hypoxemia to acute respiratory distress syndrome (ARDS). In the first 2 days of hospital admission, tachypnea, mild respiratory alkalosis and hypoxemia may occur, usually without radiological manifestations, however 33% of patients with AP have pulmonary complications with symtoms and radiological signs, some of them are atelectasis (15%), small pleural effusion (4-17%) mainly of right lung and pulmonary edema (8-50%).

Non-invasive methods would allow faster identification of patients with hypoxemia or patients who have pulmonary organ failure. (6) There is no evidence on the usefulness of SpO2 / FiO2 (SF) as a predictor of hypoxemia and its correlation with PaO2 / FiO2 in acute pancreatitis, however its continuous calculation can greatly reduce arterial gas intake and decrease adverse events and costs.

DETAILED DESCRIPTION:
Basal period

Patients will be managed based on the most current acute pancreatitis clinical guidelines and the requirements will be:

* Complete medical history including: sex, age, history of chronic degenerative diseases, pulmonary and/or cardiac diseases, alcohol consumption, onset of abdominal pain, body mass index.
* Laboratory tests: blood count, biochemical profile, amylase and serum lipase, complete serum electrolytes, lipid profile, arterial blood gases.
* Image studies:

  * Ultrasound of the upper abdomen to rule out biliary etiology
  * Computed tomography of simple abdomen in case of diagnostic doubt
  * Chest radiography
* Pulse oximetry with Finger Pulse Oximeter Brand: Carejoy Model G11002
* Severity of acute pancreatitis as follows:

  * Severity will be established based on the revised Atlanta 2012 Criteria.
  * The modified Marshall system will be evaluated to determine organic failure, which is defined as: ≥ 2 points in any of the 3 organic systems evaluated (renal, cardiovascular and pulmonary).
  * Variables will be obtained to determine systemic inflammatory response syndrome.

Intervention Arterial blood gases will be taken to calculate the PF ratio at admission and every 24 hours, until the resolution of pancreatitis and/or the first 5 days of admission.

Pulse oximetry will be performed at the same time as arterial blood gases, to calculate the SP ratio at admission and every 24 hours, until resolution of pancreatitis and/or the first 5 days of hospitalization.

Treatment The management of pancreatitis upon admission will be based on the established clinical guidelines: Hartman IV solution at 20 mL/kg and subsequently infusion at 3 mL/kg/h for the first 24 hours.

Follow up

According to the state of severity of acute pancreatitis, the following groups will be formed:

* Mild: Without multiple organic failure or ARDS
* Moderately severe or ARDS <48 hours
* Severe or ARDS> 48 hours

To assess respiratory dysfunction, 2 groups will be formed:

* No respiratory dysfunction: PF> 300
* Respiratory dysfunction: PF <300

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute pancreatitis with clinical, radiological or laboratory criteria.
* All genders
* Acute pancreatitis of any aetiology
* Over 18 years old

Exclusion Criteria:

* Lung diseases
* Heart failure
* Cholangitis
* Acute cholecystitis
* Pregnancy
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to "Dr. José Eleuterio González" University Hospital from November 2019, with diagnosis of acute pancreatitis of any etiology
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
To determine if the SpO2 / FIO2 ratio has a correlation with PaO2 / FIO2 ratio to identify respiratory compromise in acute pancreatitis. | 5 days
  Pulse oximetry will be performed at the same time as arterial blood gases, to calculate the SP ratio at admission and every 24 hours, until resolution of pancreatitis and/or the first 5 days of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda P Toalque Aldana, M.D, Principal Investigator — Hospital Univesitario
Locations (1):
- Hospital Universitario José Eleuterio González, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No